CLINICAL TRIAL: NCT02565459
Title: Third-party Bone Marrow-derived Mesenchymal Stromal Cells to Induce Tolerance in Recipients of Kidney Transplants From Deceased Donors (Phase A)
Brief Title: MSC and Kidney Transplant Tolerance (Phase A)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Monia Lorini (Other)
Collaborators: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor-Investigator, Monia Lorini, EC Secretary, A.O. Ospedale Papa Giovanni XXIII
Organization: A.O. Ospedale Papa Giovanni XXIII (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Third-party MSC-Tx tolerance A; 2015-002186-27 (EudraCT Number)
Record Dates: First submitted 2015-09-24; First posted 2015-10-01 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Chronic Renal Failure
Keywords: Mesenchymal stromal cells; kidney transplantation; tolerance
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mesenchymal Stromal Cells (MSC) (Experimental): A single intravenous infusion (1-2 millions of MSCs per kilogram body weight) of ex-vivo expanded third-party (from healthy donors) MSCs will be performed in patients randomized to the MSC procedure in addition to the kidney transplantation.
  Interventions: Biological: Mesenchymal Stromal Cells
- No intervention (No Intervention)

INTERVENTIONS:
Biological: Mesenchymal Stromal Cells
  Arms: Mesenchymal Stromal Cells (MSC)

SUMMARY:
The general aim of the present study is to test a cell therapy with third-party ex-vivo expanded bone marrow-derived mesenchymal stromal cells (MSCs) as a strategy to induce tolerance in kidney transplant recipients with a deceased donor. MSCs will be prepared accordingly to established protocols, starting from the remnants in the bag and filter at the end of the bone marrow infusions. From these samples, MSCs will be expanded in good manufacturing practice (GMP) approved facilities and used for the present study in patients undergoing kidney transplantation.

The proposed study will be developed in two phases: i) a pilot explorative safety/biologic-mechanistic phase (Phase A), ii) a pilot efficacy phase (Phase B).

ELIGIBILITY:
Inclusion Criteria:

* First single kidney transplant;
* Capable of understanding the purpose and risk of the study;
* Written informed consent.

Exclusion Criteria:

* PRA >10%;
* Specific contraindication to MSC infusion;
* Any clinical relevant condition that might affect study participation and/or study results;
* Childbearing potential without effective contraception;
* Pregnant women and nursing mothers;
* Unwillingness or inability to follow study protocol in the investigator's opinion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2015-09; Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events | Changes from baseline through study completion, up to 12 months after transplant.
  At each visit overall clinical condition of the patient will be evaluated and any adverse event will be recorded.
Circulating naive and memory T cell count (CD45RA/CD45RO) (flow cytometry analysis) | Changes from baseline at 7, 14, 30 days after transplant and then every six months through study completion, up to 12 months after transplant.
Circulating regulatory T cell count. | Changes from baseline at 7, 14, 30 days after transplant and then every six months through study completion, up to 12 months after transplant.
T-cell function in mixed lymphocyte reaction. | Changes from baseline at 6 and 12 months after transplant.
  IFNg-producing T cells (spots/300.000 cells) and CD8+ T cell-mediated cytotoxicity (percentage of specific lysis) will be measured in mixed lymphocyte reaction.
Urinary FOXP3 mRNA expression evaluated by real time quantitative PCR | Changes from baseline at 6 and 12 months after transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Remuzzi, MD, Study Chair — A.O. Ospedale Papa Giovanni XXIII; Norberto Perico, MD, Study Director — Istituto Di Ricerche Farmacologiche Mario Negri; Giovanni Rota, MD, Principal Investigator — A.O. Ospedale Papa Giovanni XXIII; Federica Casiraghi, Principal Investigator — Istituto Di Ricerche Farmacologiche Mario Negri; Martino Introna, MD, Principal Investigator — Laboratorio G. Lanzani, Bergamo, Italy; Alessandro Rambaldi, MD, Principal Investigator — A.O. Ospedale Papa Giovanni XXIII
Locations (1):
- U.O. Nefrologia e Dialisi, Bergamo, Italy